CLINICAL TRIAL: NCT02711709
Title: Persistent Inflammation, Immunosuppression and Catabolism Syndrome (PICS): A New Horizon for Surgical Critical Care Subtitle: The Acute Development and Persistence of Frailty, Comorbidity and Disability in Critically Ill Patients After Intra-abdominal Sepsis "Induced Frailty
Brief Title: Persistent Inflammation, Immunosuppression and Catabolism Syndrome (PICS): A New Horizon for Surgical Critical Care and Induced Frailty
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201501027-N; P30AG028740 (NIH)
Record Dates: First submitted 2016-02-24; First posted 2016-03-17 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
Keywords: Intra-abdominal sepsis; Surgical ICU
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intra-abdominal sepsis: Frailty measurements. Modified Minnesota Leisure Time Activities. Computed tomography morphometrics. Mobility Monitors.
  Interventions: Other: Frailty Measurements; Other: Modified Minnesota Leisure Time Activities; Other: Computed tomography morphometrics; Other: Mobility Monitors

INTERVENTIONS:
Other: Frailty Measurements — A frailty index will be determined as a combination of factors.
  An older adult is considered physically vulnerable when they experience:
  1. muscle weakness
  2. fatigue
  3. low physical activity, and unintentional loss in body weight, which has been agreed upon by a consensus of experts.
  This will be collected at baseline, 3, 6 and 12 months.
Other: Modified Minnesota Leisure Time Activities — A questionnaire used to assess physical activity will be administered at baseline, 3, 6 and 12 months.
Other: Computed tomography morphometrics — A CT scan will occur as standard of care while the patient is hospitalized. Two additional CT scans will occur at 3 and 12 months to assess for sarcopenia.
Other: Mobility Monitors — Mobility monitors will be placed on the patients during the duration of their hospital stay. They will then where them at 3, 6 and 12 months for up to 10 days.

SUMMARY:
The purpose of this study is to define the natural history and causes of chronic critical illness (CCI) in surgical intensive care patients who have had sepsis. The investigator wants to study a sub-population of sepsis patients that have intra-abdominal sepsis. The purpose of this research study is to define the acute changes in frailty (weakness, slowness, loss of muscle mass), comorbidity (medical problems) and disability (difficulty with mobility and performing routine daily functions) after having an infection that is located in the abdominal cavity or torso. The investigator believes having severe infection contributes to acute and permanent changes in these areas, especially in those of advanced age.

DETAILED DESCRIPTION:
This is a prospective study aimed at identifying the frequency, natural history and long term outcomes of CCI and PICS in the survivors of Intra-abdominal sepsis.

In addition to the in-hospital clinical data collected from the parent study, pre and post-sepsis measurements of frailty, comorbidity and disability will be obtained via questionnaires and the electronic health records. Frailty, comorbidity and disability assessments will also be completed at the three, six, and 12 month follow up assessments.

Frailty measures A frailty index will be determined as a combination of factors.

An older adult is considered physically vulnerable when they experience:

1. muscle weakness
2. fatigue
3. low physical activity, and unintentional loss in body weight, which has been agreed upon by a consensus of experts.

Two additional non-intravenous contrasted CT scans will be obtained at 3 and 12 months as part of the study protocol to assess for interval change in SMI/sarcopenia.

Objective mobility and activity monitoring will be performed to supplement assessment of frailty and disability. Wearable monitors (similar in size and appearance to a "smart watch" have received significant attention because they offer minimal burden, objectivity, versatility and low cost for assessing activity and mobility patterns. The monitor is similar in shape and size to a standard wrist watch. Thus, it will have minimal burden to patients. Each monitor will be fitted on the wrist and worn for 24 hours a day, but can be quickly removed for medical procedures, patient care or hygiene needs. Patients will wear the monitor for their entire length of stay in the hospital. It will be removed at discharge. Post-discharge, patients will be sent a monitor to wear for up to 10 days at four different time points: 3 months, 6 months and 12 months post-discharge. If study subjects are hospitalized long enough that discharge is within 30 days of the 3 month follow up, the 1 month post discharge monitoring period will be deferred. Outcomes include steps per day, total movements per day, minutes being sedentary and minutes moving at various intensities (e.g. light, moderate and vigorous).

ELIGIBILITY:
Inclusion Criteria:

* Admission to the surgery or trauma ICU where clinical care can be managed by surgical critical care guided by standard operating procedures.
* Age ≥18 years
* Diagnosis of sepsis, severe sepsis, or septic shock
* Entrance into the standard-of-care sepsis protocol
* Ability to obtain patient/legally authorized representative informed consent.

Exclusion Criteria:

* Significant traumatic brain injury (evidence of neurologic injury on CT scan and a best Glascow Coma Scale <8 within 24 hours of injury)
* Refractory shock (i.e., patients who die within 12 hours)
* Alternative or confounding diagnosis causing shock state (e.g., myocardial infarction or pulmonary embolus)
* Uncontrollable source of sepsis (e.g., irreversible disease state such as unresectable dead bowel),
* Patients deemed to be futile care or have advanced care directives limiting resuscitative efforts such as patient or patient's family who are not committed to aggressive management of the patient's condition. Expected lifespan of the patient is less than 3 months due to severe pre-existing comorbidities (ex. Recurrent, advanced or metastatic cancer).
* Severe Congestive Heart Failure (NY Heart Association Class IV)
* Child-Pugh Class C liver disease or pre-liver transplant.
* Known HIV infection with CD4 count<200 cells/mm3,
* Organ transplant recipient on immunosuppressive agents
* Known pregnancy
* Inability to obtain informed consent
* Prisoners
* Institutionalized patients
* Chemotherapy or radiotherapy within 30 days prior to sepsis
* Spinal cord injuries resulting in permanent sensory and/or motor deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intra-Abdominal Sepsis Patients
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
A change in rate of participants (0-100%) that meet frailty consensus criteria comparing baseline score to assessments after (3, 6, 12 months) episode of intra-abdominal sepsis using the Fried Frailty Criteria. | Baseline, 3, 6 and 12 months.
  1. Fried Frailty Criteria: Possible score of 0-5 based on clinical criteria. Score of 0 = "Not Frail", Score of 1-2 = "pre-frail", score ≥3 = "Frail". Integer score, no units of measures
A change in rate of participants (0-100%) that meet frailty consensus criteria comparing baseline score to assessments after (3, 6, 12 months) episode of intra-abdominal sepsis using the Rockwood Frailty Criteria. | Baseline, 3, 6 and 12 months.
  Rockwood Frailty Criteria: Ratio (0-1.0) based on number of positive clinical factors of a 70 item list of clinical deficits (i.e. 7/70 deficits = 0.1). Ratio score, no units of measure.

SECONDARY OUTCOMES:
Change in measurement of torso sarcopenia. | Baseline, 3, 6 and 12 months.
  Sarcopenia as measured by computed tomography morphometric analysis calculation of skeletal muscle index (SMI) at the level of the 3rd lumbar vertebra at baseline as compared to 3 and 6 months after intra-abdominal sepsis. Sarcopenia is defined as SMI ≤38.5 cm2/m2 for men and ≤52.4 cm2/m2.
A change in the Modified Minnesota leisure time activities questionnaire from baseline to the one year mark. | Baseline, 3, 6 and 12 month
  This measures leisure time (both free time and domestic chores) for the 2 weeks prior to the hospitalization and at each of the above referenced time points. The raw scores are indexed to a key of activity and intensity codes, which are then utilized to calculate an Activity Metabolic Index. A healthy AMI will have an intensity code of 6.0 while a fight AMI will have intensity codes of 4.0 or less.
A change in mobility and activity from hospitalization to the one year mark. | Baseline, 3, 6 and 12 months.
  This is measured as total movements per day (integer, no units of measure) and steps per day (integer, no units of measure) by portable actigraphy monitors as measured during inpatient hospitalization as compared to 1-week assessments at 3, 6 and 12 months after intra-abdominal sepsis. These measurements will be aggregated and then classified by an overall intensity index (light, moderate, vigorous).
Mortality | Up to one year
  Mortality will be assessed daily while the subject is in the hospital and then at post discharge follow up visits or by phone if the subject is unable to come to the follow up appointments. The Social Security mortality database will be accessed for subjects that are lost to follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Efron, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health at Shands hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No